CLINICAL TRIAL: NCT05243836
Title: Contact Lenses Utilising S.T.O.P.® Technology Versus Dual-focus Contact Lenses for Slowing Down Myopia Progression in Children: A Three-year Prospective, Multi-centre, Controlled, Masked, Randomised, Non Inferiority Clinical Trial
Brief Title: S.T.O.P.® Technology Contact Lenses Versus Dual-focus Contact Lenses for Slowing Down Myopia Progression in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: nthalmic Pty Ltd (Network)
Collaborators: Brighten Optix Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: nthal2021-01
Record Dates: First submitted 2022-01-17; First posted 2022-02-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MiSight® (Active Comparator): MiSight® Contact Lens (Omafilcon A, 60% water)
  Interventions: Device: MiSight®
- S.T.O.P® F2 (Experimental): S.T.O.P® F2 Contact Lens (Ocufilcon D, 55% water)
  Interventions: Device: S.T.O.P® F2
- S.T.O.P® DT (Experimental): S.T.O.P® DT Contact Lens (Ocufilcon D, 55% water)
  Interventions: Device: S.T.O.P® DT

INTERVENTIONS:
Device: S.T.O.P® F2 — Ocufilcon D, 55% water
  Arms: S.T.O.P® F2
Device: S.T.O.P® DT — Ocufilcon D, 55% water
  Arms: S.T.O.P® DT
Device: MiSight® — Omafilcon A (60% water)
  Arms: MiSight®

SUMMARY:
To compare the rate of myopia progression of contact lenses utilising S.T.O.P.® technology against MiSight® contact lenses.

DETAILED DESCRIPTION:
Myopic children (8-14 years of age) will be randomly allocated to wear one of 3 contact lens options (MiSight®, S.T.O.P.®- F2 or S.T.O.P.®- DT) bilaterally on a daily wear basis. The overall trial duration, including follow-up period, is expected to be approximately 48 months. Each participant's duration is expected to be approximately 36 months.

The visits are Baseline / Fit, Dispensing, 1 week, 1 month, 6 months then visits every 6 months after.

All procedures performed at these visits are standard, non invasive clinical tests.

ELIGIBILITY:
Inclusion Criteria:

* Be between 8-14.
* Have:

  * Read the Informed Assent.
  * Been explained the Informed Assent.
  * Indicated an understanding of the Informed Assent.
  * Signed the Informed Assent.
* Have their parent / legal guardian:

  * Read the Informed Consent.
  * Been explained the Informed Consent.
  * Indicated an understanding of the Informed Consent.
  * Signed the Informed Consent.
* Along with their parent / legal guardian, be capable of comprehending the nature of the study, and be willing and able to adhere to study requirements.
* Along with their parent / legal guardian, agree to maintain the visit schedule .
* Agree to wear allocated contact lenses for a minimum of 5 days per week, at least 6 hours per day on days lenses are worn but not > 16 hours per day, and to remove lenses at night (i.e., daily wear only with no contact lens wear during sleep), for their duration of the study and to inform the investigator if their schedule is interrupted. Wearing time can be modified by the investigator for health reasons.
* Possess wearable and visually functioning spectacles.
* Be in good general health, based on the parent's / legal guardian's knowledge.
* Have best-corrected high contrast visual acuity based on manifest refraction of 0.10 logMAR (20/25, 6/7.6) or better in each eye.
* Meet the following criteria determined by cycloplegic autorefraction:

  * Spherical equivalent between -0.75 to -4.00 D inclusive.
  * Astigmatism ≥ -1.00 D.

    *participants who fail astigmatism criterion with autorefraction pass astigmatism criterion if ≥ -0.75 D is measured with subjective refraction.
  * anisometropia ≤ 1.00 D.

Exclusion Criteria:

* Participant is currently, or within 30 days prior to this study, has been an active participant in another study.
* Current or prior use of ANY form of myopia control, including but not limited to:

  * Optical devices.

    * Bifocal / multifocal spectacles of any type.
    * Bifocal / multifocal contact lenses of any type.
    * Orthokeratology of any type.
  * Pharmacological agents.

    * European and Indian sites: Atropine.
    * Chinese sites: Atropine with a concentration > 0.01%. Participants who have previously used 0.01% atropine are eligible for this study provided they agree not to use 0.01% atropine for at least 30 days before baseline and at any time during the study.
    * Pirenzepine.
* Participant born earlier than 30 weeks or weighed < 1500 g at birth.
* Habitual use of a systemic or topical medication that may alter normal ocular findings / is known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and / or during the clinical trial.
* A known allergy to sodium fluorescein, benoxinate, proparacaine, or tropicamide.
* Chinese sites: A known allergy to cyclopentolate.
* A known corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections, or any other recurrent ocular infections.
* Strabismus by cover test at distance (3 m) or near (40 cm) while wearing distance correction under non-cycloplegic conditions.
* Known ocular or systemic disease, such as but not limited to:

  * Diabetes.
  * Graves' disease.
  * Glaucoma.
  * Uveitis.
  * Scleritis.
  * Auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjogrens syndrome, and systemic lupus erythematosus.
* Any ocular, systemic, or neuro-developmental conditions that could influence refractive development, such as but not limited to:

  * Persistent pupillary membrane.
  * Vitreous haemorrhage.
  * Cataract.
  * Central corneal scarring.
  * Eyelid haemangiomas.
  * Marfan's syndrome.
  * Down's syndrome.
  * Ehler's-Danlos syndrome.
  * Stickler's syndrome.
  * Ocular albinism.
  * Retinopathy of prematurity.
* Keratoconus or irregular cornea.
* Biomicroscopic that contraindicate contact lens, such as but limited to:

  * Neovascularisation or ghost vessels ≥ 1.5 mm in from limbus.
  * Any active anterior segment disease that contraindicates safe contact lens wear.
  * Clinically significant giant papillary conjunctivitis.
  * Clinically significant abnormalities of the anterior segment, lids, conjunctiva, sclera, or associated structures.
  * Allergic or seasonal conjunctivitis if the investigator believes it could significantly interfere with maintaining a specified wearing schedule.
* The investigator may, at their discretion, exclude anyone who they believe may not be able to fulfil the clinical trial requirements or it is believed to be in the participant's best interests.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 441 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Axial Length | Baseline, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Difference in change from baseline in axial length between test and control contact lenses.

SECONDARY OUTCOMES:
Cycloplegic spherical equivalent autorefraction | Baseline, 12 months, 24 months, 36 months
  Difference in change from baseline in spherical equivalent autorefraction between test and control contact lenses.
Visual performance as measured by high contrast visual acuity at 6 m | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in visual performance between test and control contact lenses
Visual performance as measured by a non validated questionnaire based on a 1-10 numeric rating scale where a higher score indicates a better outcome | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in visual performance between test and control contact lenses
Bulbar hyperemia graded on a 0-4 scale in 0.5- steps where a higher grading indicates increased hyperemia | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in bulbar hyperemia grading between test and control contact lenses.
Limbal hyperemia graded on a 0-4 scale in 0.5- steps where a higher grading indicates increased hyperemia | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in limbal hyperemia grading between test and control contact lenses.
Palpebral roughness graded on a 0-4 scale in 0.5- steps where a higher grading indicates increased roughness | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in palpebral roughness grading between test and control contact lenses.
Corneal staining graded on a 0-4 scale in 0.5- steps where a higher grading indicates increased staining | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in corneal staining grading between test and control contact lenses.
Conjunctival staining graded on a 0-4 scale in 0.5- steps where a higher grading indicates increased staining | 1 week, 1 month, 6 months, 12 months, 18 months , 24 months, 30 months, 36 months
  Differences in conjunctival staining grading between test and control contact lenses.
Binocular vision as measured by heterophoria in prism diopters at 3 m | 1 week, 6 months, 18 months, 30 months
  Differences in heterophoria at 3 m between test and control contact lenses.
Binocular vision as measured by heterophoria in prism diopters at 40 cm | 1 week, 6 months, 18 months, 30 months
  Differences in heterophoria at 40 cm between test and control contact lenses.
Binocular vision as measured by monocular accommodative facility (+/-2.00 D flipper) in cycles per minute at 40 cm | 1 week, 6 months, 18 months, 30 months
  Differences in monocular accommodative facility at 40 cm between test and control contact lenses.
Binocular vision as measured by monocular accommodative response in diopters at 40 cm | 1 week, 6 months, 18 months, 30 months
  Differences in monocular accommodative response at 40 cm between test and control contact lenses.
Corneal topography as measured by flat keratometry measurement in diopters | Baseline, 12 months, 36 months
  Differences in flat keratometry measurements between test and control contact lenses.
Corneal topography as measured by steep keratometry measurement in diopters | Baseline, 12 months, 36 months
  Differences in steep keratometry measurements between test and control contact lenses.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tilia, MOptom, PhD, Principal Investigator — nthalmic Pty Ltd
Locations (8):
- China (3):
  - Wenzhou Medical University Eye Hospital, Wenzhou, Lucheng District
  - Tianjin Medical University, Tianjin, Wuqing District
  - Shanghai Fudan University Eye and ENT Hospital, Shanghai, Xuhui District
- India (2):
  - LV Prasad Eye Institute, Hyderabad, Telangana
  - The University of Hyderabad, Hyderabad, Telangana
- Spain (3):
  - Centre Universitari de la Visió, Terrassa, Barcelona
  - Lab. de Superficie Ocular y Lentes de Contacto (SOYLC), Santiago de Compostela, Galicia
  - Ocupharm Research Group (Clinica Universitaria de Optometría), Universidad Complutense Madrid, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.